CLINICAL TRIAL: NCT02266342
Title: Evaluation on the Treatment of Diseases of the Thoracic Aorta With the Thoracic Endoprosthesis GORE® TAG®
Brief Title: GORE® TAG® Thoracic Endoprosthesis French Mandatory Registry
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: FPR12-03
Record Dates: First submitted 2014-10-10; First posted 2014-10-17 (Estimated); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-11

CONDITIONS: Aortic Aneurysm, Thoracic; Descending Thoracic Aortic Dissection; Aortic Diseases; Aorta Thoracic; Traumatic Rupture; Penetrating Ulcer
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Dissection, Thoracic Aorta; Aortic Diseases; Penetrating Atherosclerotic Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: GORE® TAG® Thoracic Endoprostheses — Endovascular therapy to treat thoracic disease
  Other Names: Conformable GORE® TAG® Thoracic Endoprostheses

SUMMARY:
This is a French Registry mandated by the French National Health Authority assessing long-term (5-years) safety of the GORE® TAG® Thoracic Endoprosthesis treating diseases of the thoracic aorta.

DETAILED DESCRIPTION:
Endovascular therapy to treat thoracic disease seems to provide a plausible benefit compared to surgery in terms of operative mortality and severe morbidity. The French National Health Authority (HAS) requires a 5-year follow-up as part of the renewal of reimbursement for these endoprostheses in order to collect long-term follow-up data under real-life conditions of use.

ELIGIBILITY:
Inclusion Criteria:

* Patient where a GORE® TAG® or Conformable GORE® TAG® Thoracic Endoprosthesis is implanted (successfully or not) for the treatment of disease of the descending thoracic aorta.
* Patient who had previously consented to the collection and processing of personal medical data.
* Patient older than 18 years at the time of treatment.

Exclusion Criteria:

* Patients who have already received treatment with a thoracic endoprosthesis other than the GORE® TAG® or Conformable GORE® TAG® Thoracic Endoprosthesis and for whom 'revision' or reintervention is required.
* Patients whose clinical follow-up is not possible (i.e. patients who cannot return for control visits because they live abroad).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a disease of the descending thoracic aorta, requiring treatment with a thoracic endoprosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Chakfé, Prof, Principal Investigator — Hôpitaux Universitaire de Strasbourg
Locations (1):
- Hopitaux Universitaire de Strasbourg, Strasbourg, France

RESULTS

PARTICIPANT FLOW:
Groups:
- GORE® TAG® Thoracic Endoprothesis: Patients receiving a GORE® TAG® or Conformable GORE® TAG® Thoracic Endoprosthesis implant for the treatment of a descending thoracic aortic disease.
Period: Overall Study
Arm/Group | GORE® TAG® Thoracic Endoprothesis
Started | 154
Completed | 60
Not Completed | 94

BASELINE CHARACTERISTICS:
Arm/Group | GORE® TAG® Thoracic Endoprothesis
Number analyzed (Participants) | 154
Age, Continuous [Median (Full Range); unit: years] | 68 [59 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 105
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 154
Main Indication for Implantation [Count of Participants; unit: Participants]
  Thoracic Aortic Aneurysm | 56
  Type B Dissection of the Thoracic Aorta | 60
  Traumatic Wound | 15
  Penetrating Aortic Ulcer | 17
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With All-cause Mortality (Long-term)
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® TAG® Thoracic Endoprothesis
Number analyzed (Participants) | 154
Participants | 31

2. Secondary Outcome: Number of Subjects With Excluded Aneurysm, Penetrating Aortic Ulcer (PAU), False Lumen or Site of Rupture
Time Frame: 5 years
Population: Subjects with known exclusion status at 5 years with the following main indications for implantation: Thoracic Aortic Aneurysm, Type B Dissection of the Thoracic Aorta, Traumatic Wound, or Penetrating Aortic Ulcer
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® TAG® Thoracic Endoprothesis
Number analyzed (Participants) | 64
Participants | 50

3. Secondary Outcome: Number of Subjects With Neurological Complications
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® TAG® Thoracic Endoprothesis
Number analyzed (Participants) | 154
Participants | 13

4. Secondary Outcome: Number of Subjects With Cardiac, Renal, and Pulmonary Complications
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® TAG® Thoracic Endoprothesis
Number analyzed (Participants) | 154
Participants | 32

5. Secondary Outcome: Number of Subjects With Device-related Complications
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® TAG® Thoracic Endoprothesis
Number analyzed (Participants) | 154
Participants | 8

6. Secondary Outcome: Number of Subjects With Surgical Conversion
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® TAG® Thoracic Endoprothesis
Number analyzed (Participants) | 154
Participants | 0

7. Secondary Outcome: Number of Subjects With Secondary Procedures
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® TAG® Thoracic Endoprothesis
Number analyzed (Participants) | 154
Participants | 27

8. Secondary Outcome: Number of Subjects With Disease Related Mortality
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® TAG® Thoracic Endoprothesis
Number analyzed (Participants) | 154
Participants | 5

ADVERSE EVENTS:
Time Frame: Five year follow-up
Groups:
- GORE® TAG® Thoracic Endoprothesis: GORE® TAG® and Conformable GORE® TAG® Thoracic Endoprosthesis Registiry conducted for reimbursement in France and no MedDRA coding was required.
Arm/Group | GORE® TAG® Thoracic Endoprothesis
All-Cause Mortality (participants affected / at risk) | 31/154
Serious Adverse Events (participants affected / at risk) | 79/154
Other Adverse Events (participants affected / at risk) | 38/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GORE® TAG® Thoracic Endoprothesis (N=154)
Cardiac (Cardiac disorders) | 13
Neurological (Nervous system disorders) | 12
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 12
Renal (Renal and urinary disorders) | 6
Vascular (Vascular disorders) | 40
Other (General disorders) | 24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GORE® TAG® Thoracic Endoprothesis (N=154)
Vascular (Vascular disorders) | 24
Cardiac (Cardiac disorders) | 5
Neurological (Nervous system disorders) | 2
Renal (Renal and urinary disorders) | 2
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 4
Other (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT02266342/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT02266342/SAP_001.pdf